CLINICAL TRIAL: NCT06618066
Title: Decision-making Preferences and Its Related Factors on Parents With Children Having Cancer
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-E(II)-20230162
Record Dates: First submitted 2024-08-18; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-08

CONDITIONS: Pediatric Cancer
Keywords: Decision making preferences; Parents; Coping behaviors; Family cohesion
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional correlational study was conducted in the pediatric hematology-oncology ward and outpatient clinic of a medical center in southern Taiwan. Participants included fathers or mothers of children diagnosed with cancer aged between 20 and 65 years. Structured questionnaires were used, including FACES IV, JCS, and CPS-P. This study aims to explore the current status of family cohesion, coping behaviors, and decision making preferences among parents of children with cancer, and to identify factors influencing decision making preferences.

ELIGIBILITY:
Inclusion Criteria:

1. Parents aged between 20 and 65 years whose child has been diagnosed with pediatric cancer by a physician.
2. Individuals who understand Mandarin or Taiwanese Hokkien and are able to complete the questionnaire.
3. Individuals who consent to participate in the study after being informed of the research purpose.

Exclusion Criteria:

(1)Individuals diagnosed with a mental illness by a physician.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study was conducted in the pediatric hematology-oncology ward and outpatient clinic of a medical center in southern Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Exploring the current state of decision-making preferences among parents of children with cancer using the Control Preferences Scale for Pediatrics (CPS-P) | Single point in time: At enrollment
  The CPS-P is a method for assessing individual preferences in medical decision-making roles, consisting of five options that represent five different roles.(A) I prefer to make the final decision about which treatment my child will receive, (B) I prefer to make the final selection of my child's treatment after seriously considering my doctor's opinion, (C) I prefer that my child's doctor and I share responsibility for deciding which treatment is best for my child, (D) I prefer that my doctor makes the final decision about which treatment will be used, but seriously considers my opinion, (E) I prefer to leave all decisions regarding my child's treatment to my doctor. The five responses are classified into three categories representing active(A and B), collaborative (C) and passive (D and E) decision-making preference.
Exploring the current state of family cohesion among parents of children with cancer using the Family Adaptability and Cohesion Evaluation Scale (FACES) | Single point in time: At enrollment
  The evaluation of family functioning involves: (1) Balanced Scales: Cohesion and Flexibility, (2) Unbalanced Scales: Disengaged, Enmeshed, Rigid, and Chaotic, (3) Family Communication, and (4) Family Satisfaction. The instrument consists of eight subscales with a total of 62 items, rated on a five-point Likert scale. The Family Cohesion and Flexibility scales include 42 items (0-42), divided into six sections with scores ranging from 7 to 35 per section. The Family Communication scale, which assesses positive communication and openness, contains 10 items (43-52) with scores ranging from 10 to 50. The Family Satisfaction scale, measuring satisfaction with cohesion, flexibility, and communication, also has 10 items (53-62), scoring from 10 to 50. Higher scores on Cohesion and Flexibility suggest a healthier family system; higher scores on Disengaged, Enmeshed, Rigid, and Chaotic indicate dysfunction; higher scores on Communication and Satisfaction denote more positive perceptions.
Exploring the current coping behaviors of parents of children with cancer using the Jalowiec Coping Scale (JCS) | Single point in time: At enrollment
  The Jalowiec Coping Scale (JCS) assesses eight types of coping strategies, which are categorized into emotion-oriented and problem-oriented approaches. The emotion-oriented strategies include: evasive strategies (13 items), optimistic strategies (9 items), fatalistic strategies (4 items), emotive strategies (5 items), and palliative strategies (7 items). The problem-oriented strategies include: confrontive strategies (10 items), supportant strategies (5 items), and self-reliant strategies (7 items). It utilizes a four-point Likert scale, where "0 = never used," "1 = seldom used," "2 = sometimes used," and "3 = often used." Higher scores indicate a higher frequency of coping strategy use.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Min Wu, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olson D. FACES IV and the Circumplex Model: validation study. J Marital Fam Ther. 2011 Jan;37(1):64-80. doi: 10.1111/j.1752-0606.2009.00175.x. PMID 21198689
- [Background] Degner LF, Sloan JA, Venkatesh P. The Control Preferences Scale. Can J Nurs Res. 1997 Fall;29(3):21-43. PMID 9505581
- [Background] Jalowiec A, Murphy SP, Powers MJ. Psychometric assessment of the Jalowiec Coping Scale. Nurs Res. 1984 May-Jun;33(3):157-61. PMID 6563533